CLINICAL TRIAL: NCT00535951
Title: A Phase IB, Open-Label, Multicenter Study to Investigate the Effect of Oral LBH589 on Dextromethorphan, a CYP2D6 Substrate, and to Assess the Efficacy and Safety of Oral LBH589 in Patients With Advanced Solid Tumors
Brief Title: Pharmacokinetic, Safety, and Efficacy Effects of Oral LBH589 on Dextromethorphan in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer or Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2109
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Mesothelioma
Keywords: Non-small cell lung cancer; NSCLC; lung cancer; pleural mesothelioma; malignant; advanced stage; mesothelioma; phase I; LBH589; dextromethorphan; CYP2D6; oral
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma; Lung Neoplasms; Mesothelioma, Malignant | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589

SUMMARY:
This study will investigate the effect of oral LBH589 on dextromethorphan, a CYP2D6 substrate, and to assess safety and efficacy of oral LBH589 when used with this co-medication in advanced stage NSCLC or malignant pleural mesothelioma patients

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years
2. Must have histologically or cytologically confirmed advanced or metastatic incurable solid tumor as documented by CT or MRI that has progressed on or following standard therapies
3. Must have failed prior standard systemic therapy
4. Must have at least one measurable and/or non-measurable lesion as defined by RECIST criteria
5. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal.
6. Written informed consent obtained prior to any screening procedures
7. Willingness to have multiple blood draws
8. Ability to swallow capsules or tablets

Exclusion criteria:

1. Uncontrolled brain metastases
2. Prior treatment with an HDAC inhibitor
3. Presence of clinically detectable third-space fluid collections (e.g., ascites or pleural effusions) that can not be controlled by drainage or other procedures prior to study entry
4. Concomitant use of any anti-cancer therapy, including radiation therapy
5. Significant cardiac disease
6. Concomitant use of drugs with a risk of causing torsades de pointes
7. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
8. Previous use of monoamine oxidase inhibitors (e.g. clorgyline, iproniazid, isocarboxazid, moclobemide, sibutramine, phenelzine, tranylcypromine) within 14 days prior to the first dose of dextromethorphan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters | first 10 days

SECONDARY OUTCOMES:
Response rate assessed by comparing tumor size via radiology scans (CTs or MRIs) | day 10 through end of treatment
Safety (until disease progression, unacceptable toxicity or study completion) assessed by duration of patient participation | first 10 days, day 10 through end of treatment plus follow-up
Tolerability (until disease progression, unacceptable toxicity or study completion) assessed by duration of patient participation | day 10 through end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (5):
- United States (4):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Medical College of Georgia, Augusta, Georgia
  - RUSH Medical Center, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Ontario, Canada

REFERENCES:
- See also: Results for CLBH589B2109 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2855